CLINICAL TRIAL: NCT06571175
Title: Myocardial Fibrosis With High Frame Rate Echocardiography in Patients With Aortic Stenosis - A Follow-up Study
Brief Title: Quantification of Myocardial Fibrosis in Aortis Stenosis
Acronym: SAS-F-5
Status: Enrolling by invitation | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Oslo University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 527717
Record Dates: First submitted 2024-07-10; First posted 2024-08-26 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Aortic Valve Stenosis; Myocardial Fibrosis
Keywords: High frame rate echocardiography; Heart failure; Aortic stenosis; Cardiac MRI; Prognosis; Quantification of severity
MeSH Terms: conditions — Aortic Valve Stenosis; Heart Failure | interventions — Hematologic Tests; Electrocardiography, Ambulatory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Aortic stenosis: Mild aortic stenosis:25 patients were included at baseline, and those that still avoid exclusion criteria, will be invited to undergo repeat echocardiography, MRI, blood test, questionnaires, 6 min walking test, ECG and Holter-ECG.
  Moderate aortic stenosis: 25 patients were included at baseline, and those that still avoid exclusion criteria, will be invited to undergo repeat echocardiography, MRI, blood test, questionnaires, 6 min walking test, ECG and Holter-ECG.
  Severe aortic stenosis: 50 patients were included at baseline, and those that still avoid exclusion criteria, will be invited to undergo repeat echocardiography, MRI, blood test, questionnaires, 6 min walking test, ECG and Holter-ECG.
  Interventions: Diagnostic Test: High frame rate echocardiography; Diagnostic Test: MRI; Diagnostic Test: Blood test; Diagnostic Test: ECG and Holter-ECG; Diagnostic Test: 6 min walking test
- Controls: The controls from baseline inclusion will be invited to undergo repeat echocardiography, blood test and CMRI
  Interventions: Diagnostic Test: High frame rate echocardiography; Diagnostic Test: MRI; Diagnostic Test: Blood test

INTERVENTIONS:
Diagnostic Test: High frame rate echocardiography — Conventional transthoracic echocardiography will be performed, with added 3D-imaging and acquisitions with high frame rate. The data from these patients will be anonymized and transferred for post-hoc analysis in dedicated computer software (GE Vingmed, EchoPac 2.6) and in validated machine learning algorithms.
  Other Names: GE Vingmed ultrasound scanner E95, 2017
Diagnostic Test: MRI — Cardiac MRI will be performed. In all patients without contraindications, a gadolinium-based contrast agent will be given.
  Other Names: Cardiac magnetic resonance imaging (CMRI)
Diagnostic Test: Blood test — Conventional brachial venous blood samples will be drawn. Hematocrit value {in %} will be used to calculate CMR-derived exttracellular volume (ECV)
Diagnostic Test: ECG and Holter-ECG — ECG/Holter-ECG will be performed, and the findings will be related to the imaging findings.
  Groups: Aortic stenosis
Diagnostic Test: 6 min walking test — 6 MWT will be performed, and the findings will be related to findings from CMRI/echocardiography.
  Groups: Aortic stenosis

SUMMARY:
This study is a long term follow-up of patients that were included as part of a previous study (NCT03422770), where patients with aortic stenosis and healthy controls went through echocardiography, cardiac MRI, long-term ECG-recording, blood tests and quality of life assessment. Echocardiography included high frame ultrasound for detection of natural mechanical waves, and the measured speed of these waves were used as a marker of the extent of myocardial fibrosis.

Up to five years have now passed since inclusion at baseline, and a proportion of the patients in the cohort have undergone aortic valve replacement at some point. In this study, the investigators will repeat the cardiac imaging (echocardiography and cardiac MRI), ECG and blood test, to assess long-term changes in myocardial fibrosis in aortic stenosis patients.

DETAILED DESCRIPTION:
High frame rate ultrasound with quantification of myocardial mechanical wave velocities provides a new approach to evaluation of myocardial stiffness.

Principle: An elastic medium (the left ventricle) is incited by a force (naturally occuring mechanical wave generated by atrial contraction and/or closure of mitral and aortic valve), and the resulting oscillation wave propagates through the medium with a speed that depends only on the density and stiffness of the medium. If the density of the medium is known, measuring the propagation velocity of the wave is the same as measuring the stiffness of the medium.

There is a lack of longitudinal data in this research area. A follow-up study of the described cohort, will add valuable insight into high frame rate ultrasound as a potential tool to quantify myocardial fibrosis in heart failure patient, and to monitor any changes from baseline.

ELIGIBILITY:
Inclusion Criteria:

* Part of the initial cohort that were included in the baseline study
* Still able to undergo protocolled investigations
* Patients: Mild, moderate or severe AS

Exclusion Criteria:

* Renal insufficiency
* Previously myocardial infarction (ECG, echocardiogram or hospital record)
* Severe valvular heart disease (except patients)
* Other cardiac disease known to cause myocardial fibrosis
* Severe hypertension
* Other medical conditions deterring protocolled investigation and follow-up
* Other medical conditions affecting 5-years prognosis (cancer, pulmonary disease)
* Severely reduced image-quality (echocardiography and MRI)

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients: Mild, moderate, or severe aortic valve stenosis. A subset of the patients will have undergone aortic valve replacement since inclusion.
  Controls: Healthy with no valve disease, or other cardiac disease known to cause myocardial fibrosis
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular morbidity | 5 year
  Admissions with heart failure
Cardiovascular mortality | 5 year
  Death caused by cardiac disease

SECONDARY OUTCOMES:
All cause mortality | 5 years
  Mortality in general
Time of first re-hospitalization | 5 years
  Time of first re-hospitalization after inclusion
Cardiac systolic function | 5 years
  Systolic function based on left ventricular ejection fraction (LVEF) and global longitudinal strain (GLS).
  Unit of measure for LVEF and for GLS is % for both (a positive number for LVEF, and a negative number for GLS)
Cardiac diastolic function (1 of 5) | 5 years
  Echocardiographic diastolic function based on i) left atrial volume index {ml/m^2).
Cardiac diastolic function (2 of 5) | 5 years
  Echocardiographic diastolic function based on ii) mitral annular velocities {cm/sec}
Cardiac diastolic function (3 of 5) | 5 years
  Echocardiographic diastolic function based on iii) mitral inflow velocities {cm/sec}
Cardiac diastolic function (4 of 5) | 5 years
  Echocardiographic diastolic function based on iv) ricuspid regurgitation velocity {cm/sec}
Cardiac diastolic function (5 of 5) | 5 years
  Echocardiographic diastolic function based on v) E/è-ratio
Velocity of natural mechanical waves propagating through the myocardium | 5 years
  Investigate for prognotisc value and if it can be a marker of diastolic dysfunction. Unit of velocity measurement is m/sec.

CONTACTS AND LOCATIONS:
Overall Officials: Brage H: Amundsen, MD, PhD, Principal Investigator — Norwegian University of Science and Technology (NTNU)
Locations (1):
- St. Olavs Hosptial, Trondheim, Trøndelag, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Salles S, Espeland T, Molares A, Aase SA, Hammer TA, Stoylen A, Aakhus S, Lovstakken L, Torp H. 3D Myocardial Mechanical Wave Measurements: Toward In Vivo 3D Myocardial Elasticity Mapping. JACC Cardiovasc Imaging. 2021 Aug;14(8):1495-1505. doi: 10.1016/j.jcmg.2020.05.037. Epub 2020 Aug 26. PMID 32861651
- [Background] M. Mohajery, S. Salles, T. Espeland, S. Fadnes and L. Lovstakken,
- [Result] Espeland T, Wigen MS, Dalen H, Berg EAR, Hammer TA, Salles S, Lovstakken L, Amundsen BH, Aakhus S. Mechanical Wave Velocities in Left Ventricular Walls in Healthy Subjects and Patients With Aortic Stenosis. JACC Cardiovasc Imaging. 2024 Feb;17(2):111-124. doi: 10.1016/j.jcmg.2023.07.009. Epub 2023 Sep 6. PMID 37676209